CLINICAL TRIAL: NCT00201318
Title: A Randomized Study of Lamivudine Prophylaxis or Treatment Against Hepatitis B Reactivation in Non-Hodgkin's Lymphoma Patients Carrying Hepatitis B Surface Antigen
Brief Title: A Randomized Study in Non-Hodgkin's Lymphoma Patients Carrying Hepatitis B Surface Antigen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); National Cheng-Kung University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chi Mei Medical Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1401
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: Cyclophosphamide Doxorubicin Vincristine Lamivudine

SUMMARY:
* AIMS OF THE STUDY (STUDY OBJECTIVES)

1. To test the effect of daily lamivudine (100 mg) in reducing the risk of HBV reactivation and hepatitis development in HBsAg (+) NHL patients.
2. To test the efficacy of daily lamivudine in preventing and treating hepatitis B reactivation and in circumventing hepatic failure and death.
3. To test whether lamivudine can improve the overall outcome of NHL patients who are HBV carriers.

(Study end-points: The major end-point: hepatitis B reactivation in NHL patients---defined by higher than 10-fold increase of serum HBV DNA level and/or reappearance of HBeAg in the serum during and within 6 months after chemotherapy. The minor end-point I : events of hepatic failure and death---defined by jaundice with hepatic encephalopathy. The minor end-point II: the response rate and survival rate in HBsAg-positive NHL patients receiving lamivudine prophylaxis and treatment.)

DETAILED DESCRIPTION:
* TREATMENT PLANS

  1. Systemic chemotherapy with CHOP regimen Schedule and Dose for CHOP Cyclophosphamide 750 mg/m2 i.v. Day 1 Doxorubicin 50 mg/m2 i.v. Day 1 Vincristine 1.4 mg/m2/d i.v. Day 1 Prednisolone 60 mg/m2/d p.o. Day 1-7 1.1 Courses will be repeated every 21 days. 1.2 For patients with CR, give at least 2 additional courses for a minimum of 6 courses.

     1.3 For patients with maximal response as PR or SD, change to second-line chemotherapy. The regimens for second-line chemotherapy are at the discretion of the investigators. Local radiotherapy is allowed for residual localized 1.4 For patients with PD, change to second-line chemotherapy. The regimens of the latter are at the discretion of the investigators.

     2.1 Arm I Patients take lamivudine 100 mg P.O. qd, starting from Day 1 of the first course of CHOP, and until 2 months after the completion of chemotherapy. Lamivudine is to be maintained no matter hepatitis occurred or not during chemotherapy. If second-line chemotherapy is used, lamivudine with the same dose and schedule will be continued until 2 months after completion of the second-line chemotherapy.

     If third-line chemotherapy is needed, the use of lamivudine will be at the 2.2 Arm II Patients are treated with CHOP alone. If the patients develop clinical hepatitis, as defined in section 7.2, lamivudine 100 mg, P.O., qd., will be given, and continued until hepatitis is resolved. Prophylactic lamivudine is not to be given in subsequent chemotherapy. (Our previous study has indicated that nearly all clinical hepatitis developed in HBV carriers during systemic chemotherapy is caused by HBV reactivation. Therefore, for practical reason, the investigators are not advised to wait for the results of HBV DNA serology examination before starting lamivudine treatment. )

     3.0 DOSE MODIFICATION 3.1 Hematological Toxicity* Drug administration is postponed if there is no full hematological recovery (AGC > 2,000/mm3 and Platelet > 100,000/mm3 ) from prior course at scheduled treatment day. Full doses will be given as soon as the hematological recovery is documented. If two weeks after the due day recovery is still incomplete, the treatment may be started and the dosage be reduced according to the following

     schedule:

     AGC*/mm3Platelet/mm3 1,500-2,00075,000-100,000 1,000-1,49950,000-74,999 <1,000<50,000 Cyclophosphamide 80% 60% ** Doxorubicin 80% 60% **
* G-CSF is allowed to be used prophylactically for older ( > 60 years old) patients and for patients with previous or ongoing prolonged myelosuppression.

  * Postpone for another week. If the counts remain AGC<1,500 or Platelet <75,000 three weeks after the due day, patients should be off study.

3.2 Hepatotoxicity For patients with normal prechemotherapy serum ALT, hepatitis flare-up is defined as ALT elevation greater than 1.5 fold of upper normal limit. For patients with abnormal prechemotherapy serum ALT, hepatitis flare-up is defined as 2.0 fold or greater increase of serum ALT level. The hepatitis or hepatitis flare-up is attributed to reactivation of HBV when there is a sudden elevation (>10-fold) in serum HBV DNA level or reappearance of HBV DNA and/or HBeAg in the serum.

Since results of our previous study has indicated that nearly all clinical hepatitis developed in HBV carrier during chemotherapy is caused by HBV reactivation, and serum HBV DNA data are not readily available in most hospitals, all patients with hepatitis flare-up are considered HBV reactivation until proved otherwise. For patients in the second arm, biochemical hepatitis will prompt a start of daily lamivudine, even before a definite documentation of 10-fold increase of HBV DNA. For patients with only minor hepatic dysfunction (total bilirubin <3.0 mg/dl and ALT <200 I.U./L), full-dose chemotherapy is recommended on the scheduled treatment day without delay. For patients with more severe hepatic dysfunction (total bilirubin ≧ 3.0 mg/dl or ALT ≧ 200 I.U./L), subsequent course is postponed for 1 week and the dosage modified as followings if the values remain abnormal after 1 week:

Total Bilirubin (mg/dl) <3.0 3.0 ~ 4.9 5.0 ~ 7.5 >7.5 ALT (I.U./L) <200 200 ~ 399 400 ~ 800 >800 Doxorubicin 100% 75% 50% *

* Wait until recovery with serum levels below these values. Patients will be off study if Bil > 7.5 mg/dl or ALT > 800 I.U/L, 3 weeks after the due day.

3.3 Gastrointestinal Toxicity In case of severe (≧ NCI Gr III) anorexia, nausea, vomiting, diarrhea, stomatitis or abdominal pain, all therapy should be delayed until improvement of symptoms to ≦ GrII.

Patients will be off study if ≧ Gr III toxicity persists ≧ 3 weeks after due day. Patients are allowed to use H3-blockers in the subsequent courses for severe nausea and vomiting. If gastrointestinal toxicity is still ≧ Gr III during the next course, doses of cyclophosphamide and doxorubicin should be reduced by 25% in the subsequent courses. If no further episodes of severe reaction, the doses can be escalated, 12.5% each time, and back to 100%.

3.4 Cardiotoxicity In case of NCI grade II cardiotoxicity, doxorubicin should be reduced by 50%. If cardiotoxicity is resolved, the dose may be carefully deescalated, 12,5% each time, in the subsequent courses. If severe (≧ NCI grade III) cardiotoxicity develops, doxorubicin should be discontinued and should not be used again in the subsequent courses.

3.5 Multiple Toxicity In the event of multiple toxicity, dose modification should be based on the guideline that requires the greatest reduction of doses.

4.0 CRITERIA FOR REMOVAL FROM STUDY

All patients who are still under or have completed protocol treatments (1st-line or 2nd-line) should be continuously followed-up for all study end points. Patients are removed from study if they have major violation of the protocol due to the following reasons:

1. Completion of assigned therapy and observation.
2. Progressive of disease.
3. Excessive of complication or toxicity.
4. Patient death.
5. Patient withdrawal or refusal.

5.0 MEASUREMENT OF EFFECT ： Authorized physicians or research nurses must call Ms. Yueh-Ling Ho at the TCOG Operations Office (Tel: 02-26534401 ext 6655) for patients registration and randomization.

A permuted block randomization will be used to generate the list by the Statistical Center housed at the Division of Biostatistics, NHRI. Treatment assignment is given only when the patient passes the eligibility check.

6.0 REPORT OF ADVERSE EFFECT : Adverse effect of treatments should be reported to TCOG Operations Office at 02-26534401 ext 6655, 6657, 6658 and FAX: 02-2782-3755, within 48 hours. See appendix for the TCOG ADR (Adverse Drug Reaction) Form of reporting adverse effect.

ELIGIBILITY:
* Inclusion Criteria:

  1. Histologically proven NHL, and for which intensive chemotherapy is considered treatment-of-choice.
  2. HBsAg-positive.
  3. No previous chemotherapy and radiotherapy, no concurrent radiotherapy.
  4. AGC ≧ 2,000/mm3, Platelet ≧ 100,000/mm3 of peripheral blood.
  5. Total bilirubin < 2.5 mg/dl. Alanine aminotransferase (SGPT) < 200 I.U./L
  6. Serum creatinine ≦1.5 mg/dl Blood urea nitrogen (BUN) ≦ 25 mg/dl
  7. Objectively measurable or valuable disease
  8. Signed informed consent
* Exclusion Criteria:

  1. Age > 75 years old, or Age < 15 years old
  2. Pregnant or breast-feeding women.
  3. Patients with history of brain metastasis or CNS involvement.
  4. Child's class B or C in patients with liver cirrhosis.
  5. Impaired cardiac function with NYHA (New York Heart Association) classification ≧ Gr II.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-09; Study Completion 2005-10

PRIMARY OUTCOMES:
We expect to enter 33 patients per year. Taking into account 10﹪dropout rate, we may finish accrual of patients within 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, Ph.D., Study Chair — National Taiwan University Hospital; Ann-Lii Cheng, Ph.D., Study Chair — National Taiwan University Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan